CLINICAL TRIAL: NCT05692986
Title: Randomized Control Trial: Chlorhexidine vs Povidone Iodine Vaginal Prep in Decreasing Postoperative Infection in Total Laparoscopic Hysterectomy
Brief Title: Chlorhexidine vs Povidone Iodine Vaginal Prep in Decreasing Postoperative Infection in Total Laparoscopic Hysterectomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Did not move forward due to staffing
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Joelle Abood, Principal Investigator, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 15037
Record Dates: First submitted 2022-01-23; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Preventative Laparoscopic Hysterectomy
Keywords: 4% chlorhexidine; 10% povidone iodine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- povidone betadine (Active Comparator)
  Interventions: Diagnostic Test: A vaginal swab for aerobic and anaerobic cultures before antibiotic administration, 30 minutes after vaginal prep and every hour thereafter until the surgery is completed.
- chlorhexidine (Active Comparator)
  Interventions: Diagnostic Test: A vaginal swab for aerobic and anaerobic cultures before antibiotic administration, 30 minutes after vaginal prep and every hour thereafter until the surgery is completed.

INTERVENTIONS:
Diagnostic Test: A vaginal swab for aerobic and anaerobic cultures before antibiotic administration, 30 minutes after vaginal prep and every hour thereafter until the surgery is completed. — This is a randomized control trial that will compare chlorhexidine vaginal prep with iodine vaginal prep. Our primary outcome will be assessed using a vaginal swab test to look for aerobic and anaerobic cultures. Positive cultures will be defined as colony forming count of >5000cfu. All patients will receive preoperative antibiotics. Patients will receive a vaginal swab for aerobic and anaerobic cultures before antibiotic administration, 30 minutes after vaginal prep and every hour thereafter until the surgery was completed.

SUMMARY:
This is a randomized control trial which will randomize patients who will be undergoing laparoscopic (conventional or robotic assisted) total hysterectomy to vaginal prep with 4% chlorhexidine gluconate vs 10% povidone iodine. There is paucity of information regarding the superiority of one over the other.

DETAILED DESCRIPTION:
This is a randomized control trial. During surgery, preoperative vaginal prep is routinely done for hysterectomies. This can be completed with 10% povidone iodine or with 4% chlorhexidine preparation. This study will investigate whether the routine use of betadine vaginal prep in comparison to chlorhexidine prep is superior. Patients will be informed of the study at the time of their preoperative visit in the gynecology clinic at time of surgical scheduling. The attached informed consent sheet will be given to the patient for their signature. The patients will be randomized to receive either 10% povidone iodine or with 4% chlorhexidine vaginal preparation solution. This is not anticipated to take extra time or resources in the operating room setting because the surgical vaginal preparation solutions are typically readily available in the operating room setting. The patients will be assigned an envelope when they are in clinic after they have signed the consent form and that will be the group they are randomized to.

Once the patients are randomized, it is anticipated that 50 patients will be enrolled in each study arm. Following randomization patients will receive the vaginal preparation per the randomization assignment. The patient will be blinded to the study arm. The provider will not be blinded. Follow-up will occur on postoperative day #1 by phone call, and at the 2-week and 6-week follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled for total laparoscopic hysterectomy

Exclusion Criteria:

* not able to consent in English or have allergy to the 10% povidone betadine or 4% chlorhexidine solution.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
The number of positive cultures in each arm will be compared. | before antibiotic administration, 30 minutes after vaginal prep and q1hr thereafter until the surgery was completed
  The number of positive cultures in each arm will be assessed using vaginal swabs to look for contaminated specimens. Positive cultures will be defined as colony forming counts of >5000cfu, and these will be compared in each arm to determine which preparation is more effective

IPD SHARING:
Plan to Share IPD: No